CLINICAL TRIAL: NCT06463587
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled, 3-Arm, 3-Period Study to Assess the Efficacy and Safety of a New Formulation of Oral Cladribine Compared With Placebo in Participants With Generalized Myasthenia Gravis (MyClad)
Brief Title: Efficacy and Safety of a New Formulation of Oral Cladribine Compared With Placebo in Participants With Generalized Myasthenia Gravis (MyClad)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: EMD Serono Research & Development Institute, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MS700568_0183; 2023-507746-83-00 (Other: EU CTIS)
Record Dates: First submitted 2024-06-11; First posted 2024-06-18 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Generalized Myasthenia Gravis
Keywords: Anti-AChR antibody positive; anti-MuSK antibody positive; anti-LRP4 antibody positive; seronegative gMG
MeSH Terms: conditions — Myasthenia Gravis | interventions — Cladribine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): DBPC Period: Participants will be administered with Placebo, orally as 2 separate treatment courses starting on Day 1 and at the beginning of Week 5.
  BE Period: Participants initially randomized to placebo matched to cladribine in DBPC period will receive cladribine Low Dose or High Dose, orally as 2 separate treatment courses starting at the beginning of Week 25 and at the beginning of Week 29 and retreated if clinically justified with placebo matched to cladribine.
  RT Period: Participants requiring retreatment with cladribine Low Dose or High Dose or retreated with cladribine supplemental dose if clinically justified.
  Interventions: Other: Placebo; Drug: Cladribine Low Dose; Drug: Cladribine High Dose
- Cladribine Low Dose (Experimental): DBPC Period: Participants will be administered with cladribine Low Dose, orally as 2 separate treatment courses starting on Day 1 and at the beginning of Week 5.
  BE Period: Participants initially randomized to cladribine Low Dose in DBPC period will receive placebo matched to cladribine as 2 separate treatment courses starting at the beginning of Week 25 and at the beginning of Week 29 and retreated with cladribine supplemental dose if clinically justified.
  RT Period: Participants requiring retreatment with cladribine Low Dose regimen and/or supplemental dose will receive the selected dose of cladribine if clinically justified.
  Interventions: Drug: Cladribine Low Dose
- Cladribine High Dose (Experimental): DBPC Period: Participants will be administered cladribine High Dose, orally as 2 separate treatment courses starting on Day 1 and at the beginning of Week 5.
  BE Period: Participants initially randomized to cladribine High Dose in DBPC period will receive placebo matched to cladribine as 2 separate treatment courses starting at the beginning of Week 25 and at the beginning of Week 29 and retreated with cladribine supplemental dose if clinically justified.
  RT Period: Participants requiring retreatment with cladribine High Dose regimen and/or supplemental dose will receive the selected dose of cladribine if clinically justified.
  Interventions: Drug: Cladribine High Dose

INTERVENTIONS:
Other: Placebo — Participants will receive placebo matched to cladribine in two courses separated by 4 weeks.
  Arms: Placebo
Drug: Cladribine Low Dose — Participants will receive cladribine low dose in two courses separated by 4 weeks.
  Arms: Cladribine Low Dose; Placebo
Drug: Cladribine High Dose — Participants will receive cladribine high dose in two courses separated by 4 weeks.
  Arms: Cladribine High Dose; Placebo

SUMMARY:
The purpose of this clinical study is to determine the efficacy and safety of a new oral cladribine formulation in participants with Generalized Myasthenia Gravis (gMG) in comparison to placebo. It will also investigate the sustained efficacy, the need for retreatment, and the long-term safety of oral cladribine in gMG. An additional component is included to characterize the Pharmacokinetics (PK) of the new cladribine formulation in gMG participants. This study is divided into 3 periods: the double-blind placebo control (DBPC) pivotal period, and 2 extensions, the blinded extension (BE) and the retreatment (RT) period.

ELIGIBILITY:
Inclusion Criteria:

* Adults of ≥ 18 years of age at the time of signing the informed consent.
* Diagnosis of Myasthenia Gravis with generalized muscle weakness, meeting clinical criteria for Myasthenia Gravis Foundation of America Class II to IVa classification.

  * In participants positive for Acetylcholine receptor antibody (anti-AChR) or muscle-specific kinase antibody(anti-MuSK)
  * In participants that are autoantibody seronegative and participants who are positive for anti-low-density lipoprotein receptor-related protein 4 antibodies (anti-LRP4)
* Has a Screening and Baseline MG-ADL score more than or equal to (>=) 6 with >= 50 percentage (%) of the total score due to non-ocular symptoms. Screening and Baseline MG-ADL scores must be stable. The difference between the Screening and Baseline scores should not be more than 2 and there should be no reported MG exacerbation during the Screening period
* If treated with oral corticosteroids: should be on a stable daily dose for at least 3 months prior to and during screening. In such case, the daily dose of oral steroids should not exceed 20 milligrams(mg)/day for prednisone/ prednisolone or 16 mg/day for methylprednisolone
* If treated with acetylcholinesterase inhibitor should be on a stable daily dose (pyridostigmine dose ≤ 480 mg/day) for at least 3 months prior to and during screening
* Have a body weight >= 40 kilograms
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Immunologic disorder other than MG or any other condition requiring chronic oral, intravenous, intramuscular, or intraarticular corticosteroid therapy. Well-controlled thyroid disease, as per the Treating Investigator or the participants regular treating physician recorded in the source documents, is not exclusionary
* Molecularly characterized or suspected congenital myasthenic syndrome, Lambert-Eaton myasthenic syndrome, inherited myopathy, muscular dystrophy, acquired myopathy or any other neurologic or systematic disease that mimics MG muscular weakness
* Active, clinically significant viral, bacterial, or fungal infection, including brain MRI findings consistent with signs of infection such as PML, or any major episode of infection requiring hospitalization or treatment with parenteral anti-infectives within 8 weeks prior or during Screening, or completion of oral anti-infectives within 8 weeks prior or during Screening. Vaginal candidiasis, onychomycosis, and genital or oral herpes simplex virus considered by the Investigator to be sufficiently controlled would not be exclusionary
* Has a history of or current diagnosis of active tuberculosis (TB)
* Active malignancy, or history of cancer
* Treatment with nonsteroidal immunosuppressants, used in gMG, such as azathioprine, mycophenolate mofetil, methotrexate, cyclosporine, tacrolimus within 4 weeks prior to randomization
* Treatment with eculizumab, rozanolixizumab efgartigimod, ravulizumab, or zilucoplan within 8 weeks prior to randomization
* History of thymectomy within 6 months prior to Screening.
* History of generalized seizures (except for history of infantile febrile seizures)
* Negative for Varicella Zoster Virus antibodies at screening
* History of myasthenic crisis in the last 12 months prior to and during screening
* History of recurrent infections (that is 3 or more infections per year) within the last 2 years
* Discontinuation of treatment with any non-steroidal immunosuppressants used in gMG, such as azathioprine, mycophenolate mofetil, methotrexate, cyclosporine, tacrolimus within the last 6 months prior to Screening
* If treated with non-steroidal immunosuppressants for gMG, the dose at Screening should not exceed 50 mg/day for azathioprine, 500 mg/day for mycophenolate mofetil, 1 mg/day for tacrolimus, 50 mg/day for cyclosporine, or 7.5 mg/week for methotrexate
* Participation in clinical study of any investigational drug within 6 months, or 5 half-lives of the investigational drug used in the previous clinical study prior to randomization, whichever is longer. However, participants with any prior exposure to cladribine may not enter the study regardless of timing of exposure
* Other protocol defined exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2024-06-25 (Actual); Primary Completion 2028-05-19 (Estimated); Study Completion 2030-08-19 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Myasthenia Gravis - Activities of Daily Living (MG-ADL) Scale Score at Week 24 During the Double-Blind Placebo Controlled (DBPC) Period | Baseline, Week 24

SECONDARY OUTCOMES:
Change from Baseline in Quantitative Myasthenia Gravis (QMG) Scale Score at Week 24 During the Double-Blind Placebo Controlled (DBPC) Period | Baseline, Week 24
Percentage of MG-ADL Responders at Week 24 During the Double-Blind Placebo Controlled (DBPC) Period | At Week 24
  MG-ADL responder is defined by achieving >= 3 points decrease in MG-ADL score.
Change from Baseline in Myasthenia Gravis Composite (MGC) Scale Score at Week 24 During the Double-Blind Placebo Controlled (DBPC) Period | Baseline, Week 24
Percentage of Quantitative Myasthenia Gravis (QMG) Scale Responders at Week 24 During the Double-Blind Placebo Controlled (DBPC) Period | At Week 24
  QMG responder is defined by achieving >= 4 points decrease in QMG score.
Time From Initial Cladribine Full Dose Treatment to First Retreatment or Rescue Treatment up to end of Study | Up to End of Study (Week 144)
Number of Participants With Adverse Events (AEs) and Adverse Events of Special Interest (AESIs) | Up to End of Study (Week 144)
Number of participants with Adverse Events (AEs) by Severity as per National Cancer Institute Common Terminology Criteria for Adverse Events, version 5.0 | Up to End of Study (Week 144)
Number of Participants with Abnormal Laboratory Variables including Absolute Lymphocyte Count and Vital Signs | Up to End of Study (Week 144)
Pharmacokinetic (PK) Plasma Concentration of Cladribine | Pre-dose, 0.25, 1, 2, 3, 4, 6, 8 and 24 hours post-dose
Change from Baseline in the Revised Myasthenia Gravis Quality of Life - 15 Scale (MG-Qol15r) Score at Week 24 During the Double-Blind Placebo Controlled (DBPC) Period | Baseline, Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — EMD Serono Research & Development Institute, Inc.
Locations (112):
- United States (17):
  - Arizona Neuroscience Research, LLC, Phoenix, Arizona
  - Advanced Neurosciences Research LLC, Longmont, Colorado
  - The George Washington University Medical Faculty Associates Foggy Bottom South Pavilion, Washington D.C., District of Columbia
  - Neurology of Central Florida Research Center, LLC, Altamonte Springs, Florida
  - SFM Clinical Research, LLC, Boca Raton, Florida
  - University of Florida Health Science Center - 300120311, Jacksonville, Florida
  - Neurology Associates, P. A., Maitland, Florida
  - University of South Florida - PARENT - PARENT, Tampa, Florida
  - University of Kansas Medical Center Research Institute, Inc. - 3901 Rainbow (MAIN), Kansas City, Kansas
  - Atrium Health Wake Forest Baptist, Winston-Salem, North Carolina
  - Miami Valley Hospital South, Centerville, Ohio
  - Clinical Trials of South Carolina - Charleston, Charleston, South Carolina
  - Erlanger Health, Inc. - 1123255, Chattanooga, Tennessee
  - Baylor Scott & White Research Institute - Baylor Scott & White Research Institute, Dallas, Texas
  - ANESC Research, El Paso, Texas
  - The University of Vermont Medical Center, Burlington, Vermont
  - Integrated Neurology Services - Dr. Simon Fishman's Office, Falls Church, Virginia
- Argentina (8):
  - Expertia S.A- Mautalen Salud e Investigación, Ciudad Autonoma Buenos Aires
  - Instituto de Investigaciones Neurologicas Raul Carrea, FLENI - de Investigaciones Clinicas del área de Cardiología y enfermedades metabólicas asociadas, Ciudad Autonoma Buenos Aires
  - Instituto de Investigaciones Metabolicas (IDIM), Ciudad Autonoma Buenos Aires
  - Hospital Cordoba, Córdoba
  - Fundacion Rosarina de Neurorehabilitacion, Rosario
  - INECO Neurociencias Oroño, Rosario
  - CER San Juan Centro Polivalente de Asistencia e Inv. Clinica, San Juan
  - Centro de Investigaciones Medicas Tucuman, San Miguel de Tucumán
- Australia (3):
  - Sunshine Coast University Hospital, Birtinya, Queensland
  - Box Hill Hospital - PARENT, Box Hill, Victoria
  - Gold Coast University Hospital - PARENT, Southport
- Belgium (2):
  - UZ Leuven, Leuven
  - C. H. R. de la Citadelle - Account 1, Liège
- Bulgaria (5):
  - Medical Center Hera - branch Montana, Montana
  - UMHAT 'Dr. Georgi Stranski', EAD, Pleven
  - UMHAT "Sv. Georgi", EAD, Plovdiv
  - MHATNP "Sv.Naum", EAD - Third Neurology Clinic, Sofia
  - UMHATEM 'N.I. Pirogov', EAD, Sofia
- China (15):
  - The First Affiliated Hospital of Bengbu Medical College, Anhui Sheng, Anhui
  - Xuanwu Hospital Capital Medical University, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Guangzhou University of Chinese Medicine - 300164595, Guangzhou, Guangdong
  - Affiliated Hospital of Zunyi Medical University, Zunyi, Guizhou
  - Shijiazhuang People's Hospital, Shijiazhuang, Hebei
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Xiangya Hospital, Central South University, Changsha, Hu'nan
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science & Technology, Wuhan, Hubei
  - The First Hospital of Jilin University - The First Hospital of Jilin University, Changchun, Jilin
  - China-Japan Union Hospital of Jilin University - 300173736, Changchun, Jilin
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Huashan Hospital, Fudan University - Neurology, Shanghai, Shanghai Municipality
  - Xi 'an International Medical Center, Xi’an, Shanxi
  - West China Hospital, Sichuan University, Chengdu, Sichuan
- France (5):
  - CHU de Grenoble - Hôpital Albert Michallon - Centre de Références des Maladies Neuromusculaires, La Tronche, Isere
  - CHU Clermont Ferrand - Hopital Gabriel Montpied - service de neurologie B, Clermont-Ferrand, Puy De Dome
  - Hopital Neurologique Pierre Wertheimer - Pathologies neuro-musculaires. Electromyographie, Bron, Rhone
  - Hôpital Henri Mondor - Service de Neurologie, Créteil, Val De Marne
  - Groupe Hospitalier Pitie-Salpetriere - Centre Référent Maladies Rares SLA - Neurologie, Paris
- Georgia (3):
  - Ltd. Pineo Medical Ecosystem, Tbilisi
  - New Hospitals LLC, Tbilisi
  - Aversi Clinic Ltd, Tbilisi
- Germany (4):
  - Medizinische Hochschule Hannover - Klinik fur Neurologie mit Klinischer Neurophysiol, Hanover, Lower Saxony
  - St. Joseph Hospital - St. Joseph Hospital Haan, Bochum, North Rhine-Westphalia
  - Universitaetsklinikum Carl Gustav Carus TU Dresden - Medizinische Klinik I, Dresden, Saxony
  - Charité Universitaetsmedizin Berlin - Campus Charité Mitte - Klinik fuer Neurologie, Berlin
- University Hospital of Patra, Pátrai, Greece
- India (7):
  - Nizam's Institute of Medical Sciences, Hyderabad, Andhra Pradesh
  - Yashoda Super Speciality Hospital - 300158817, Hyderabad, Andhra Pradesh
  - Bangalore Medical College and Victoria Hospital - 300148268, Bangalore, Karnataka
  - St John's Medical College Hospital, Bangalore, Karnataka
  - Mallikatta Neurocentre, Mangalore, Karnataka
  - Chopda Medicare & Research Centre - 300188248, Nashik, Maharashtra
  - Deenanath Mangeshkar Hospital and Research Centre - Department of Neurology, Pune, Maharashtra
- Italy (4):
  - Policlinico Universitario Agostino Gemelli - UOC Neurologia, Rome, Roma
  - Azienda Socio Sanitaria Territoriale Papa Giovanni, Bergamo
  - IRCCS Ospedale Policlinico San Martino - Neuroradiologia, Genova
  - Fondazione Istituto Neurologico Casimiro Mondino - Neurology, Pavia
- Japan (11):
  - Chiba University Hospital - Dept of Neurology, Chiba, Chiba
  - IUHW Narita Hospital - Dept of Neurology, Narita-shi, Chiba
  - Southern Tohoku Medical Clinic - Dept of Neurology, Koriyama-shi, Fukushima
  - Hakodate Municipal Hospital - Dept of Neurology, Hakodate-shi, Hokkaido
  - General Hanamaki Hospital - Dept of Neurology, Hanamaki-shi, Iwate
  - Kagawa University Hospital - Dept of Neurology, Kita-gun, Kagawa-ken
  - Nagasaki University Hospital - Dept of Neurology, Nagasaki, Nagasaki
  - Saitama Medical University Hospital - Dept of Neurology/Stroke Care Unit, Iruma-gun, Saitama
  - Toho University Ohashi Medical Center - Dept of Neurology, Meguro-ku, Tokyo-To
  - Tokyo Medical University Hospital - Dept of Neurology, Shinjuku-ku, Tokyo-To
  - Osaka University Hospital - Dept of Neurology/Stroke Care Unit, Suita-shi
- Poland (4):
  - Uniwersyteckie Centrum Kliniczne - Dept of Neurology, Gdansk
  - Krakowska Akademia Neurologii Sp z o.o. Centrum Neurologii Klinicznej, Krakow
  - MTZ Clinical Research Powered By Pratia, Warsaw
  - Wielospecjalistyczne Centrum Medyczne Ibismed - Dept of Neurology, Zabrze
- Romania (2):
  - S.C Neurocity S.R.L, Bucharest
  - Spitalul Clinic Judetean de Urgenta Targu Mures - Sectia Clinica Neurologie I, Târgu Mureş
- South Korea (7):
  - Kyungpook National University Chilgok Hospital, Daegu
  - Chonnam National University Hospital, Gwangju
  - Samsung Medical Center, Seoul
  - Korea University Anam Hospital, Seoul
  - Asan Medical Center, Seoul
  - Seoul Metropolitan Government Seoul National University Boramae Medical Center, Seoul
  - Keimyung University Dongsan Hospital, Seoul
- Spain (5):
  - Hospital Universitari Germans Trias i Pujol - Servicio de Neurologia, Badalona, Barcelona
  - Hospital Universitario Reina Sofia - Neurology Dept, Córdoba, CÃ³rdoba
  - Hospital Universitario Central de Asturias - Servicio de Neurologia, Oviedo, Principality of Asturias
  - Hospital Universitari Vall d'Hebron - Neurology Dept, Barcelona
  - Hospital Universitari i Politecnic La Fe - Pediatry Department, Valencia
- Sweden (3):
  - Sahlgrenska Sjukhuset, GÃ¶teborg
  - Centralsjukhuset Karlstad, Karlstad
  - Danderyd Sjukhus - 300147691, Stockholm
- Taiwan (4):
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Shin Kong Wu Ho-Su Memorial Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- United Kingdom (2):
  - Nottingham University Hospitals NHS Trust, Nottingham, Nottinghamshire
  - Royal Hallamshire Hospital - Dept of Neurology, Sheffield, South Yorkshire

IPD SHARING:
Plan to Share IPD: Yes
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website bit.ly/IPD21
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Within six months after the approval of a new product or a new indication for an approved product in both the United States and the European Union
Access Criteria: Qualified scientific and medical researchers can request the data. Such requests must be submitted in writing to the company's portal and will be internally reviewed regarding criteria for researchers' qualification and legitimacy of the research proposal.
URL: http://bit.ly/IPD21

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS700568_0183
- See also: US Medical Information website, Medical Resources — https://medical.emdserono.com/en_US/home.html
- See also: Related Info — http://www.mycladstudy.com